CLINICAL TRIAL: NCT06615245
Title: A Magic Bowl Low Tech Vs. High Tech Immersive Virtual Reality Distraction
Brief Title: Measuring Attention During Immersive Virtual Reality Distraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Hoffman (Other)
Responsible Party: Sponsor-Investigator, Hunter Hoffman, Director, Principle Investigator, Sr. Research Scientist, University of Washington
Organization: University of Washington (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UWashington
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-09

CONDITIONS: Distraction
Keywords: virtual reality; distraction

STUDY DESIGN:
Intervention Model Description: within subject repeated measures design with treatment order randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant will eventually get to try virtual reality, but participants will not be informed that some people receive a more immersive virtual reality than other people. In other words, participants will remain blind to the high tech vs. Low tech VR manipulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- n = 16 participants: No VR condition vs. Immersive VR (Sham Comparator): Participants will perform a simple attention demanding task during No VR for 2 minutes, and again during a Immersive High Tech Virtual Reality game distraction. They will also rate how distracted they were and how hard it was to concentrate on the attention demanding task during each 2 minute task.
  Interventions: Behavioral: No VR vs. immersive high tech VR
- n = 20 participants: plausible control (see through VR) condition vs. immersive High Tech VR (Active Comparator): 20 healthy volunteer participants will perform a simple attention demanding task during a plausible control (see through) VR for 2 minutes, and again during an immersive High Tech Virtual Reality distraction (treatment order randomized). They will also rate how distracted they were and how hard it was to concentrate on the attention demanding task during the 2 minute tasks. During Phase 2 they will also rate their pain and anxiety during a brief thermal stimulus Quantitative Sensory Testing) during No VR vs. during immersive High Tech VR.
  Interventions: Behavioral: Plausible control vs immersive High Tech VR

INTERVENTIONS:
Behavioral: No VR vs. immersive high tech VR — No VR vs. immersive High Tech VR
  Arms: n = 16 participants: No VR condition vs. Immersive VR
Behavioral: Plausible control vs immersive High Tech VR — plausible control condition vs. immersive high tech VR
  Arms: n = 20 participants: plausible control (see through VR) condition vs. immersive High Tech VR

SUMMARY:
Brief Summary

Using a repeated measures within-subject design with treatment order randomized, with healthy volunteers, this study will measure how much immersive Virtual Reality (VR) reduces performance on a simple attention demanding task during No VR vs. High Tech VR (for one group of 16 participants), and during a plausible control see through VR vs. High Tech VR (for another group of 20 participants).

The primary aim is to explore whether a highly immersive VR system makes VR significantly more attention demanding/distracting, compared to No VR, and compared to a less immersive VR system (a plausible controlled see through goggles).

DETAILED DESCRIPTION:
Healthy college student volunteers will participate in a repeated measure within subject trial studying attention using a divided attention paradigm.

One group of participants (16 healthy volunteers) will perform a simple attention demanding task during No VR for 2 minutes and they will perform the attention demanding task again during High Tech VR for 2 minutes.

Another group of 20 healthy volunteers will perform a simple attention demanding task during a less immersive see through VR (a plausible control condition) for 2 minutes and they will also perform the attention demanding task again during immersive High Tech VR for 2 minutes (treatment order randomized). This group will also rate their pain and anxiety during Quantitative Sensory Testing very brief thermal heat stimuli during No VR vs. during immersive high tech VR.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a course at the University of Washington Psychology Dept., participating in the University of Washington (UW) Psychology subject pool
* Able to read, write and comprehend English
* Able to complete study measures
* Willing to follow our UW approved instructions
* 18 years of age or older

Exclusion Criteria:

* People who have already previously participated in this same study (e.g., last quarter) are not eligible to participate again.
* Not enrolled in a course at the University of Washington Psychology Dept., not participating in the UW Psychology subject pool
* Not be able to read, write and comprehend English
* Younger than 18 years of age.
* Not capable of completing measures
* Not capable of indicating pain intensity,
* Not capable of filling out study measures,
* Extreme susceptibility to motion sickness,
* Seizure history,
* Unusual sensitivity or lack of sensitivity to pain,
* Sensitive skin,
* Sensitive feet
* Migraines
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
accuracy on an attention demanding cognitive test | for n = 16, responses will be made 15 seconds after the VR condition vs. 15 seconds after the No VR during 2 minute sessions. For n = 20 subjects responses will be made 15 s after the plausible control condition, and 15 seconds after the immersive VR.
  Number of correct responses on a divided attention task

SECONDARY OUTCOMES:
graphic rating scale presence ratings | measured immediately after each two minute VR session.
  Graphic rating scale measures of patients illusion of "being there" in virtual reality.
graphic rating scale subjective pain ratings | immediately after each brief Quantitative Sensory Testing thermal heat stimulus
  n = 20 participants report how much pain they experienced during No VR vs. during High Tech VR.

OTHER OUTCOMES:
Graphic Rating Scale Difficulty performing the task and difficulty concentrating | immediately after each 2 minute session
  subjective ratings of difficulty performing the simple attention task

CONTACTS AND LOCATIONS:
Overall Officials: Hunter G Hoffman, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual data regarding participants gender, age, their accuracy on the simple attention task, and subjective ratings of difficulty performing the simple attention task, will be available upon to researchers who provide a methodologically sound proposal
Time Frame: data set and data dictionary will be available indefinitely, beginning when the paper is officially published
Access Criteria: Researchers who provide a methodologically sound proposal (e.g, for meta-analysis).